CLINICAL TRIAL: NCT07200609
Title: The Effects of a Virtual Reality-Based Gamified Rehabilitation Program on Body Structure and Function, Activity, and Participation in Children With Hemophilia: A Randomized Controlled Trial
Brief Title: The Effects of Virtual Reality-Based Gamified Rehabilitation in Children With Hemophilia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Duygu Turker, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E2-25-10575
Record Dates: First submitted 2025-09-11; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia A Without Inhibitor
Keywords: virtual reality; home-based exercise; joint health; body structure and function; activity; participation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The cases included in the study will be randomly divided into two groups using the web-based www.randomizer.org application. Group 1 is the virtual reality group, and Group 2 is the home-based exercise group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality group (Experimental): Inclusion criteria:
  Diagnosed with Hemophilia A by a pediatric hematologist Aged 6-18 years With moderate to severe hemophilia Not regularly exercising No active bleeding complaints Children who are willing to participate in the study and continue prophylactic treatment
  Exclusion criteria:
  Children with active bleeding complaints Children who have undergone lower extremity surgery Children with neurological, orthopedic, or psychological conditions that affect functional performance
  Interventions: Other: Virtual Reality Intervention
- Home-Based Exercise Group (Active Comparator): Inclusion criteria:
  Diagnosed with Hemophilia A by a pediatric hematologist Aged 6-18 years With moderate to severe hemophilia Not regularly exercising No active bleeding complaints Children who are willing to participate in the study and continue prophylactic treatment
  Exclusion criteria:
  Children with active bleeding complaints Children who have undergone lower extremity surgery Children with neurological, orthopedic, or psychological conditions that affect functional performance
  Interventions: Other: Home-Based Exercise Intervention

INTERVENTIONS:
Other: Virtual Reality Intervention — The virtual reality training group will have sessions lasting 40 minutes, 3 days a week for 8 weeks.
  * A 30-minute VR-based training session using Kinect Xbox (5 min warm-up, 30 min VR, 5 min cool-down)
  * The device has an infrared camera sensor (Kinect sensor) that detects the participant's movement in real time
  * Even if the user's movement is not performed correctly in the game settings, the user receives visual and auditory sensory feedback about movement errors.
  * All games are provided to engage participants' interest in the topics and require the use of the person's lower extremities.
  * Each game will be played for 10 minutes during the 30-minute training session. (A total of 3 games will be played)
  * Participants in VR programs typically perform active hip flexion, hip abduction, hip external and internal rotation, knee flexion and extension, ankle dorsiflexion, and plantar flexion while standing.
  * Game content: Kinect Sports, Kinect Adventures and Kinect Sports Rivals.
  Arms: Virtual reality group
Other: Home-Based Exercise Intervention — * Home-based exercise training group will also be given online exercises 3 days a week for 8 weeks.
  * Active/passive stretching exercises within pain limits
  * Patients will perform exercises at home under a supervised exercise program
  * They will perform exercises matching the virtual reality group in terms of exercise sequence, intensity, duration, and mode, incorporating open and closed kinetic chain movements
  * A 20-second stretch followed by a 20-second relaxation performed five times per session for each muscle
  * Light resistance exercises targeting muscle groups in the lower extremities, with a 5-second contraction followed by a 5-second relaxation, performed five times per session
  * Bodyweight exercises
  * Balance exercises
  * Posture exercises
  Arms: Home-Based Exercise Group

SUMMARY:
Hemophilia is an inherited bleeding disorder caused by deficiencies or low levels of clotting factors VIII (hemophilia A) and IX (hemophilia B). It is a chronic disease that negatively affects physical function, mobility, and quality of life by causing damage to joint and muscle structures due to bleeding disorders. Traditional rehabilitation methods can sometimes be boring for children and lead to a loss of motivation. Therefore, there is a need for innovative methods that will increase treatment compliance and improve children's physical activity levels.

Virtual reality (VR) technology provides a realistic and interactive environment that enables children to actively participate in the rehabilitation process. Combined with gamification elements, VR offers a fun learning and practice environment that supports the development of motor skills, reduces fear of movement, and can increase motivation for repetitive exercises.

This randomized controlled trial will evaluate the effects of virtual reality-based gamified rehabilitation on joint health, pain, posture, gait function, proprioception, and quality of life. Additionally, the contribution of this intervention to changes in activity and participation levels will be demonstrated using the International Classification of Functioning, Disability, and Health (ICF) model.

This study has the potential to guide future clinical practice by offering a more enjoyable and effective rehabilitation alternative for children with hemophilia. The widespread adoption of virtual reality-supported programs will be an important step in reducing physical disabilities associated with hemophilia.

ELIGIBILITY:
Inclusion Criteria:

* Hemophilia A diagnosed by a pediatric hematologist
* Boys aged 6-18
* Have moderate to severe hemophilia
* Do not exercise regularly
* Be able to move independently or with minimal support (ambulatory)
* Have the capacity to understand research instructions
* Prevent active bleeding
* Voluntary participation in expenses and parental record keeping
* Continued prophylactic treatment

Exclusion Criteria:

* Children with active bleeding
* Those who have had lower extremity surgery
* Those with mental retardation
* Children with neurological, orthopedic, or psychological illnesses that may affect functional performance

Ages: 6 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Hemophilia Joint Health Score (HJHS) | From enrollment to the end of treatment at 8 weeks
  HJHS is a commonly used clinical assessment scale developed to evaluate joint health in patients with hemophilia. It aims to detect hemophilia-related joint damage early, particularly in children and adolescents. Purpose of development: To detect hemophilic arthropathy (joint damage) through physical examination without the need for radiological methods. Scope: The elbow, knee, and ankle joints, which are the most commonly affected joints in hemophilia patients, are evaluated.
  Target group: Although initially developed for children aged 4-18, it is now also used in adults. The following joint characteristics are scored in the HJHS:
  Joint swelling (acute/chronic) Muscle atrophy Joint pain Loss of joint range of motion (ROM) Crepitus (sound or friction sensation during joint movement) Gait (walking) assessment Scoring: These parameters are evaluated for each joint using a specific scoring system.
  A total score of 0 = normal joint health, a higher score = more joint damage.
Physical Activity Questionnaire for Children (PAQ-C) | From enrollment to the end of treatment at 8 weeks
  Target group: Children and adolescents. Objective: To determine the level of physical activity performed through play, sports, and exercise in daily life.
  Method: The child is asked to indicate how many times they performed the activities on the list (e.g., jumping rope, running, cycling, walking, skating, games) in the last 7 days.
  Answer options:
  Never done it = 0 points 1-2 times = 1 point 3-4 times = 2 points 5-6 times = 3 points 7 times and above = 4 points Points awarded for all activities (e.g., jumping rope, running, cycling, walking, skating, tag, etc.) are added together. This total gives the child's total physical activity score for the last 7 days.
CHO-KLAT (Canadian Hemophilia Outcomes-Kids' Life Assessment Tool) | From enrollment to the end of treatment at 8 weeks
  Purpose of development: To measure the daily life experiences, social participation, and quality of life of children with hemophilia.
  Age group:
  Child version (8-18 years) → Completed by the child. Parent version (for ages 0-7 and 8-18) → Based on parental observation. Includes questions that relate conditions specific to hemophilia (e.g., bleeding, treatment burden, physical limitations) to quality of life.
  CHO-KLAT assesses the child's life from a physical, social, and emotional perspective.
  The question topics are generally:
  School and social activities (participation, friendships, involvement in games) Physical activities (sports, games, ability to exercise) Daily living activities (mobility, care, freedom of movement) Emotional state (anxiety, feelings about illness) Experiences related to treatment (injections, access to healthcare) Each item is scored between 0 and 4 (0 = strongly disagree, 4 = strongly agree).
  All scores are then added up and converted to a 0-100 range.

SECONDARY OUTCOMES:
Stability Index | From enrollment to the end of treatment at 8 weeks
  The Hur SmartBalance device is a digital system used primarily in clinical settings to assess balance, postural control, and weight transfer.
  Purpose: To objectively measure balance, detect balance disorders, and monitor the rehabilitation process.
  It includes a pressure-sensitive platform/force plate. The patient's weight distribution, sway, and stability level are recorded as numerical values.
  Both assessment and exercise can be performed thanks to the visual feedback screen.
  Parameters to be Evaluated:
  Stability Index Indicates how stable the person is in static/dynamic balance.
Posture | From enrollment to the end of treatment at 8 weeks
  The DIERS device is an advanced technology system used in clinics and research for gait analysis, posture assessment, and spinal measurements. General Features of the DIERS System Uses an optical 3D/4D scanning method → does not expose the body to radiation. It is non-invasive; there is no need to attach sensors to the child or adult. Provides detailed data on posture, spinal alignment, pressure distribution, and gait in a short time (within seconds).
  Posture and Spinal Analysis
  With the DIERS formetric (4D spine & posture) system:
  Spinal alignment (curvatures in the sagittal and frontal planes: scoliosis, kyphosis, lordosis) Shoulder and pelvic asymmetries Head and torso position Body imbalance (lateral shift, rotations) Postural balance Postural changes over time are monitored and evaluated.
Multidimensional Hemophilia Pain | From enrollment to the end of treatment at 8 weeks
  The Multidimensional Hemophilia Pain Scale (MHPQ / MHPS) is a measurement tool developed to assess the characteristics of pain in hemophilia patients in a multidimensional manner and is used in clinical practice and research. Although the MHPQ/MHPS shows minor variations across different studies, it generally covers the following areas:
  Pain intensity (severity) - typically assessed using a visual analog scale (VAS) or a 0-10 rating scale.
  Pain frequency - assessment of daily, weekly, or monthly bleeding/pain episodes.
  Pain duration - acute (minutes-hours) or chronic (weeks-months). Pain location - which joints or muscle groups are affected. Pain type - sharp, aching, throbbing, burning, etc. Functional effects of pain - impact on daily activities, sleep, school/work attendance, mobility.
  Emotional/psychosocial dimension - anxiety, depression, limited social participation.
Proprioception | From enrollment to the end of treatment at 8 weeks
  The JTECH Digital Inclinometer: This is a highly accurate digital goniometer/inclinometer that measures the angular movement of joints.
  It provides more reliable and repeatable measurements than traditional goniometers.
  The following method is used to assess proprioception (the ability to sense the position of a joint in space) in the hio and knee joints:
  Target Position Sense (JPS):
  The device is placed on the joint. The participant's joint is passively or actively moved to a specific angle (e.g., 30° of flexion for the knee).
  This angle is recorded as the reference angle.
  Target Repetition:
  The participant attempts to move the joint to the same position with their eyes closed.
  The JTECH device measures the difference between the actual angle and the target angle in degrees.
  Results:
  The smaller the margin of error, the better the proprioception. Measurements can be made separately for the hip and knee.
Functional Independence Score in Hemophilia (FISH) | From enrollment to the end of treatment at 8 weeks
  FISH is a specialized scale developed to assess functional independence in activities of daily living in patients with hemophilia. It measures the functional reflection of joint health and movement capacity in children and adults with hemophilia.
  FISH examines a total of 8 activities under 4 main categories:
  * Lower extremity movements (Leg function) Sitting down and standing up Climbing stairs Walking (on level ground)
  * Upper extremity movements (Arm function) Eating food (table setting) Wearing clothes
  * Balance/postural function Standing Bending or reaching forward
  * Fine motor skills (Fine motor function) Grasping and carrying objects Scoring
  Each activity is scored from 1 to 4:
  1. = Completely dependent
  2. = Partially dependent
  3. = Slightly dependent
  4. = Completely independent The total score is obtained by summing the activity-based scores. Higher score: Better functional independence. Lower score: More joint damage or loss of function.
Postural Sway | From enrollment to the end of treatment at 8 weeks
  The Hur SmartBalance device is a digital system used primarily in clinical settings to assess balance, postural control, and weight transfer.
  Purpose: To objectively measure balance, detect balance disorders, and monitor the rehabilitation process.
  It includes a pressure-sensitive platform/force plate. The patient's weight distribution, sway, and stability level are recorded as numerical values.
  Both assessment and exercise can be performed thanks to the visual feedback screen.
  Parameters to be Evaluated:
  Postural Sway Staying centered while standing, sway distance and speeds.
Weight Distribution | From enrollment to the end of treatment at 8 weeks
  The Hur SmartBalance device is a digital system used primarily in clinical settings to assess balance, postural control, and weight transfer.
  Purpose: To objectively measure balance, detect balance disorders, and monitor the rehabilitation process.
  It includes a pressure-sensitive platform/force plate. The patient's weight distribution, sway, and stability level are recorded as numerical values.
  Both assessment and exercise can be performed thanks to the visual feedback screen.
  Parameters to be Evaluated:
  Weight Distribution Percentage of weight transfer to the right/left, front/back.
Dynamic Balance Test | From enrollment to the end of treatment at 8 weeks
  The Hur SmartBalance device is a digital system used primarily in clinical settings to assess balance, postural control, and weight transfer.
  Purpose: To objectively measure balance, detect balance disorders, and monitor the rehabilitation process.
  It includes a pressure-sensitive platform/force plate. The patient's weight distribution, sway, and stability level are recorded as numerical values.
  Both assessment and exercise can be performed thanks to the visual feedback screen.
  Parameters to be Evaluated:
  Dynamic Balance Tests Measured by tasks such as shifting weight in specific directions and following virtual targets.
Step Length and Step Width | From enrollment to the end of treatment at 8 weeks
  The DIERS device is an advanced technology system used in clinics and research for gait analysis, posture assessment, and spinal measurements. General Features of the DIERS System Uses an optical 3D/4D scanning method → does not expose the body to radiation. It is non-invasive; there is no need to attach sensors to the child or adult. It provides detailed data on posture, spinal alignment, pressure, and gait in a short time (within seconds).
  Gait Analysis
  With DIERS' pedogait or gaitlab systems:
  Step length, step width
Cadence (Steps per Minute) | From enrollment to the end of treatment at 8 weeks
  The DIERS device is an advanced technology system used in clinics and research for gait analysis, posture assessment, and spinal measurements. General Features of the DIERS System Uses an optical 3D/4D scanning method → does not expose the body to radiation. It is non-invasive; there is no need to attach sensors to the child or adult. It provides detailed data on posture, spinal alignment, pressure, and gait in a short time (within seconds).
  Gait Analysis
  With DIERS' pedogait or gaitlab systems:
  Cadence (number of steps/min) Number of steps per minute measured with the DIERS gait analysis system. Measurement Unit: steps/minute
Right/left load distribution | From enrollment to the end of treatment at 8 weeks
  The DIERS device is an advanced technology system used in clinics and research for gait analysis, posture assessment, and spinal measurements. General Features of the DIERS System Uses an optical 3D/4D scanning method → does not expose the body to radiation. It is non-invasive; there is no need to attach sensors to the child or adult. It provides detailed data on posture, spinal alignment, pressure, and gait in a short time (within seconds).
  Gait Analysis
  With DIERS' pedogait or gaitlab systems:
  Right/left load distribution The load ratio transferred to the right and left lower extremities during walking.
  Measurement Unit: %
Pressure distribution (foot pressure patterns) | From enrollment to the end of treatment at 8 weeks
  The DIERS device is an advanced technology system used in clinics and research for gait analysis, posture assessment, and spinal measurements. General Features of the DIERS System Uses an optical 3D/4D scanning method → does not expose the body to radiation. It is non-invasive; there is no need to attach sensors to the child or adult. It provides detailed data on posture, spinal alignment, pressure, and gait in a short time (within seconds).
  Gait Analysis
  With DIERS' pedogait or gaitlab systems:
  Pressure distribution (foot pressure patterns) Pressure distribution on the sole of the foot using the DIERS pedogait system. Unit of Measurement: kPa

IPD SHARING:
Plan to Share IPD: No